CLINICAL TRIAL: NCT06724094
Title: Using Machine Learning to Detect and Predict Loosening NexGen Total Knee Replacement
Brief Title: Artificial Intelligence to Detect Early Total Knee Replacement Implant Failure
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: T&O0238
Record Dates: First submitted 2024-11-06; First posted 2024-12-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-12

CONDITIONS: Aseptic Loosening of Prosthetic Joint

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Failed: This group will be made up of patient who had revision TKR due to aseptic loosening within 10 years of primary arthroplasty
- Well performing: This group will be made up of patients who have an asymptomatic TKR 10 years after primary arthroplasty.

SUMMARY:
The goal of this trial is to investigate whether Machine Learning (ML) can be used to detect small degrees of loosening, lucent zones, or any other changes on radiographs that might predict early failure following NexGen total knee replacement.

Researchers will identify plain AP and lateral plain film radiographs from two groups of patients. Those who has NexGen total knee replacements (TKRs) that went on to failure, and those who has well performing TKRs. Radiographs from these two groups will be labelled as 'failure' and 'well performing' and will be processed through a machine learning algorithm.

The algorithm will be successful if it is able to detect a NexGen TKR that went on to failure or went on to perform well. This will be determined by using a test set.

The population will be adults who had the recalled a NexGen Total Knee Replacement with a standard tibial tray. It will include adults only, who has the TKR at University Hospitals Southampton between 2003 and 2022.

Failure will be defined as revision of tibial or femoral components which is likely due to aspectic loosening. It will exclude washouts, exchange of poly, peri-prosthetic fractures, microbiologically confirmed infection.

Well performing TKRs will be defined as patients who have had their TKR in situ for 10 years and have reported no significant symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Had a NexGen TKR between 2003 and 2022.

Exclusion Criteria:

* Below 18 yrs old.
* Revision surgery for any reason other than aseptic loosening
* patients who have not had a revision but who do not have a well functioning TKR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be adults who had the recalled a NexGen Total Knee Replacement with a standard tibial tray. It will include adults only, who has the TKR at University Hospitals Southampton between 2003 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 2105 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Predictive accuracy of machine learning model | Up to 21 years. Data starts from 2003.
  The predictive accuracy of a machine learning algorithm. Using common ML measured, AUROC etc.